CLINICAL TRIAL: NCT00640159
Title: Tolerability and Efficacy of Switch From Oral Selegiline to Orally Disintegrating Selegiline (Zelapar) in Patients With Parkinson's Disease.
Brief Title: Selegiline to Zelapar Switch Study in Parkinson Disease Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Joseph Jankovic, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-20709
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Results first posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; selegiline to Zelapar switch; orally disintegrating formulation
MeSH Terms: conditions — Parkinson Disease | interventions — Selegiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Selegiline (Experimental): Open label switch from current oral selegiline dose to orally disintegrating selegiline (Zelapar) titrated to a dose of 2.5 mg QD.
  Interventions: Drug: Zelapar

INTERVENTIONS:
Drug: Zelapar — Switch from oral selegiline to Zelapar 1.25 mg QD titrated to 2.5 mg QD
  Other Names: orally disintegrating selegiline

SUMMARY:
Parkinson's disease (PD) is a progressive neurodegenerative disease. Symptomatic therapy is primarily aimed at restoring dopamine function in the brain. Oral selegiline in conjunction with L-dopa has been a mainstay of therapy for PD patients experiencing motor fluctuations for many years. The mechanisms accounting for selegiline's beneficial adjunctive action in the treatment of PD are not fully understood. Inhibition of monoamine oxidase (MAO) type B (MAO-B) activity is generally considered to be of primary importance.

Oral selegiline has low bio-availability and is typically dosed BID, for a total of 5-10 mg daily. Recently, the FDA approved a new orally disintegration tablet (ODT) formulation of selegiline, called ZelaparTM. This new formulation utilizes Zydis technology to dissolve in the mouth, with absorption through the oral mucosa, thereby largely bypassing the gut and avoiding first pass hepatic metabolism. This allows more active drug to be delivered at a lower dose. Consequently, Zelapar is dosed once-daily, up to 2.5 mg per day. There are no empirical data indicating whether the use of the new approved formulation of selegiline ODT (Zelapar) is superior or preferred by patients compared to traditional oral selegiline. It is believed that clinical efficacy will be preserved or enhanced, by delivering more active drug, with improved patient preference for the ODT formulation due to the once-daily dosing .

The effectiveness of orally disintegrating selegiline as an adjunct to carbidopa/levodopa in the treatment of PD was established in a multicenter randomized placebo-controlled trial (n=140; 94 received orally disintegrating selegiline, 46 received placebo) of three months' duration. Patients randomized to orally disintegrating selegiline received a daily dose of 1.25 mg for the first 6 weeks and a daily dose of 2.5 mg for the last 6 weeks. Patients were all treated with levodopa and could additionally have been on dopamine agonists, anticholinergics, amantadine, or any combination of these during the trial. At 12 weeks, orally disintegrating selegiline-treated patients had an average of 2.2 hours per day less "OFF" time compared to baseline. Placebo treated patients had 0.6 hours per day less "OFF" time compared to baseline. These differences were significant (p < 0.001). Adverse events were very similar between drug and placebo.

DETAILED DESCRIPTION:
This is an open label, multicenter, 6 week study of the conversion from oral selegiline to orally disintegrating selegiline in PD patients with or without motor fluctuations, and currently taking levodopa. The study consists of the substitution of the oral selegiline with 1.25 mg of orally disintegrating selegiline for 10 days, and up titration of orally disintegrating selegiline to 2.5 mg per day for the next 30 days. The study will consist of 2 study visits in the clinic: Baseline and Day 40, and a telephone visit at Day 10.

Inclusion Criteria:

1. Idiopathic PD confirmed by at least two of the following signs: resting tremor, bradykinesia, rigidity 2. Male or female outpatients 3. Age 30-90 years 4. Current use of levodopa and oral selegiline (5-10 mg /day), stable for at least 1 month and well tolerated 5. Positive treatment response to current anti-parkinsonian medications in the opinion of the investigator 6. Acceptable contraception for females of child bearing potential 7. Willing and able to comply with study procedures. 8. Willing and able to give written informed consent prior to beginning any study procedures.

Exclusion Criteria:

1. Atypical parkinsonism due to drugs, metabolic disorders, encephalitis, trauma, or other neurodegenerative diseases. 2. Significant cognitive or psychiatric impairment which, in the opinion of the investigator, would interfere with the ability to complete all the tests required in the protocol. 3. Participation in another clinical drug trial within the previous four weeks. 4. Patients on any medications contraindicated with Zelapar (including meperidine/Demerol, tramadol, methadone, propoxyphene, dextromethorphan, other selegiline products) 5. Patients with a known hypersensitivity to any formulation of selegiline or any of the inactive ingredients of Zelapar, or previous exposure to orally disintegrating selegiline 6. History of melanoma 7. Unstable/uncontrolled medical problems 8. History of drug/alcohol abuse 9. Patients currently taking rasagiline

The primary efficacy point is number of subjects who prefer Zydis selegiline vs. the number who prefer oral selegiline, or have no preference. Descriptive statistics will be used to present the percentages of persons and adverse event resolutions. The secondary endpoints will include changes in the UPDRS, PDQ-8, BDI, FSS, ESS, ratings of global improvement and change in dyskinesia from Baseline to the Day 40 visit. Appropriate parametric (t-tests) and non-parametric analyses (Wilcoxon signed rank comparisons) will be conducted based on the scale being analyzed. An intent to treat approach will be used in which all subjects receiving at least one dose of study medication will be included in the analyses.

Tolerability and efficacy of switching from oral selegiline to Zydis selegiline in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic PD confirmed by at least two of the following signs: resting tremor, bradykinesia, rigidity
2. Male or female outpatients
3. Age 30-90 years
4. Current use of levodopa and oral selegiline (5-10 mg /day), stable for at least 1 month and well tolerated
5. Positive treatment response to current anti-parkinsonian medications in the opinion of the investigator
6. Acceptable contraception for females of child bearing potential
7. Willing and able to comply with study procedures.
8. Willing and able to give written informed consent prior to beginning any study procedures.

Exclusion Criteria:

1. Atypical parkinsonism due to drugs, metabolic disorders, encephalitis, trauma, or other neurodegenerative diseases.
2. Significant cognitive or psychiatric impairment which, in the opinion of the investigator, would interfere with the ability to complete all the tests required in the protocol.
3. Participation in another clinical drug trial within the previous four weeks.
4. Patients on any medications contraindicated with Zelapar (including meperidine/Demerol, tramadol, methadone, propoxyphene, dextromethorphan, other selegiline products)
5. Patients with a known hypersensitivity to any formulation of selegiline or any of the inactive ingredients of Zelapar, or previous exposure to orally disintegrating selegiline
6. History of melanoma
7. Unstable/uncontrolled medical problems
8. History of drug/alcohol abuse
9. Patients currently taking rasagiline

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-01; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Greg Kricorian, MD, Study Director — Valeant Pharmaceuticals
Locations (5):
- United States (5):
  - Dee Silver, MD at Coastal Neurological Medical Group, Inc, La Jolla, California
  - James Tetrud, MD at The Parkinson's Institute, Sunnyvale, California
  - Stuart Isaacson, MD at Parkinson's Disease and Movement Disorder Center of Boca Raton, Boca Raton, Florida
  - R. Malcolm Stewart, MD at Neurology Specialists of Dallas, Dallas, Texas
  - PDCMDC 6550 Fannin, Suite 1801, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ondo WG, Hunter C, Isaacson SH, Silver DE, Stewart RM, Tetrud JW, Davidson A. Tolerability and efficacy of switching from oral selegiline to Zydis selegiline in patients with Parkinson's disease. Parkinsonism Relat Disord. 2011 Feb;17(2):117-8. doi: 10.1016/j.parkreldis.2010.10.001. Epub 2010 Nov 16. PMID 21084213

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Participants received 1.25mg of orally disintegrating selegiline for 10 days, and up titration of orally disintegrating selegiline to 2.5mg per day for the next 30 days or switched from oral selegiline to Zelapar 1.25mg per day titrated to 2.5mg per day.
Period: Overall Study
Arm/Group | All Study Participants
Started | 48
Patients Who Preferred Zydis Selegiline | 25
Patients Who Preferred Oral Selegiline | 13
Patients Who Had no Specific Preferred Medication | 10
Completed | 46
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: 48 subjects were recruited. 46 subjects completed the study. 25 participated in the Zydis group, 13 participated in the Selegiline group and 10 participated in the No Preference group. 2 subjects were lost to follow-up.
Arm/Group | All Study Participants
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 34
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression Scale
Description: Baseline assessments included a clinical global impression scale. This is compared to day 40 assessment. The clinical global impression scale consists of a 3-item observer-rated scale that measures illness severity, global improvement or change and therapeutic response. Each item is rated between 1-7. The minimum score is 3. The maximum score is 21. A score of 3 means the patient's symptoms are very much improved. A score of 21 means the patient is very much worse.
Time Frame: baseline versus 40 days
Population: Clinical Global Impression scale comparison at day 40
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 48
units on a scale
  Clinical Global Impression scale at baseline | 21 (7.2)
  Clinical Global Impression scale at day 40 | 27 (4.2)

2. Secondary Outcome: MDS-UPDRS Scale at Baseline and Day 40
Description: Baseline assessment include The Movement Disorders Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS). This is compared to day 40 assessment. The MDS-UPDRS consist of 65 items. Each item can be rated between 0-4. The minimum sore is Zero. Zero means the patient is absent of Parkinson's disease symptoms. The maximum score is 260. 260 means the patient has severe Parkinson's disease symptoms.
Time Frame: baseline versus day 40
Population: MDS-UPDRS comparison at baseline and day 40
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All Study Participants: Participants received 1.25mg of orally disintegrated selegiline for 10 days, and up titration of orally disintegration selegiline to 2.5mg per day for the next 30 days or switched from oral selegiline to Zelapar 1.25mg per day titrated to 2.5mg per day.
Arm/Group | All Study Participants
Number analyzed (Participants) | 48
score on a scale
  MDS-UPDRS at baseline | 19 (3.5)
  MDS-UPDRS at day 40 | 22 (4.1)

ADVERSE EVENTS:
Time Frame: 6 week multicenter study
Groups:
- Zydis: Patients who preferred Zydis selegiline
- Selegiline: Patients who preferred oral selegiline
- No Preference: Patients who have no specific preferred medication
Arm/Group | Zydis | Selegiline | No Preference
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/13 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/13 | 0/10
Other Adverse Events (participants affected / at risk) | 3/25 | 3/13 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zydis (N=25) | Selegiline (N=13) | No Preference (N=10)
increased dyskinesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
orthostatic hypotension (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
bad taste (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
fatigue (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
fall (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
freezing (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
dry mouth (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
anxiety (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No